CLINICAL TRIAL: NCT00884442
Title: Randomized, Non-blind, 4-fold Crossover Study on Safety, Tolerability and Pharmacokinetics of Nifedipine After Single Oral Doses of Adalat® LA 60 mg or of a Marketed Generic Version of Nifedipine Retard 60 mg After an Overnight Fasting or Immediately After a High-fat American Breakfast in Healthy Male Volunteers
Brief Title: Nifedipine Bioavailability Study With Oral Single Doses Under Fasting and Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SocraTec R&D GmbH (Other)
Collaborators: SocraMetrics GmbH (Industry)
Responsible Party: Maria Anschütz, Project manager, SocraTec R&D GmbH
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 1215ni09ct
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2009-10-21 (Estimated); Status verified 2009-10

CONDITIONS: Bioavailability, Therapeutical Indication Not Studied
Keywords: Healthy; Bioavailability; Nifedipine
MeSH Terms: interventions — Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): One tablet of Gen-nifedipine extended release, previously referred to as Gen-Nifedipine XL, fasted state
  Interventions: Drug: Nifedipine (Gen-nifedipine extended release, previously referred to as Gen-Nifedipine XL)
- 2 (Active Comparator): One tablet of Gen-nifedipine extended release, previously referred to as Gen-Nifedipine XL, fed state
  Interventions: Drug: Nifedipine (Gen-nifedipine extended release, previously referred to as Gen-Nifedipine XL)
- 3 (Active Comparator): One tablet of Nifedipine (Bayer Healthcare AG manufactured as Adalat® XL®, Adalat® LA, Adalat® Crono, Adalat® OROS, fasted state
  Interventions: Drug: Nifedipine (Bayer Healthcare AG manufactured as Adalat® XL®, Adalat® LA, Adalat® Crono, Adalat® OROS)
- 4 (Active Comparator): One tablet of Nifedipine (Bayer Healthcare AG manufactured as Adalat® XL®, Adalat® LA, Adalat® Crono, Adalat® OROS, fed state
  Interventions: Drug: Nifedipine (Bayer Healthcare AG manufactured as Adalat® XL®, Adalat® LA, Adalat® Crono, Adalat® OROS)

INTERVENTIONS:
Drug: Nifedipine (Gen-nifedipine extended release, previously referred to as Gen-Nifedipine XL) — 60 mg nifedipine
  Other Names: Nifedipine 60 mg, GITS
  Arms: 1; 2
Drug: Nifedipine (Bayer Healthcare AG manufactured as Adalat® XL®, Adalat® LA, Adalat® Crono, Adalat® OROS) — 60 mg nifedipine
  Arms: 3; 4

SUMMARY:
The present study will be performed to investigate and to compare the in-vivo performance of the two investigational products Gen-nifedipine extended release, (previously referred to as Gen-Nifedipine XL (Genpharm ULC, Canada)) and Nifedipine(Bayer Healthcare AG manufactured as Adalat® XL®, Adalat® LA, Adalat® Crono, Adalat® OROS) by comparing their pharmacokinetic parameters after oral single dose administrations in the fasted and fed state.

DETAILED DESCRIPTION:
In the past, several attempts have been made to develop nifedipine formulations with pharmacokinetic characteristics similar to the unique characteristics of nifedipine GITS. A new extended release nifedipine tablet based on an osmotically active system for once a day administration has been registered under the trade name Gen-nifedipine extended release, (previously referred to as Gen-Nifedipine XL (Genpharm ULC, Canada)) in Canada.

According to the product monograph of Gen-nifedipine extended release, (previously referred to as Gen-Nifedipine XL), this tablet consists of a semipermeable membrane surrounding an osmotically active drug core. After contact with water from the GI tract osmotic pressure in the core increases, releasing the active drug at a controlled rate through an orifice in the tablet membrane. The functional principle of this nifedipine tablet seems to be quite similar to the one of the GITS system.

However, especially in case of modified release formulations, various factors can affect the absorption and the systemic availability of the drug. Two important factors are i) the drug release rate from the dosage form and ii) the gastrointestinal transit rate, which in turn has an influence on the site of absorption. Especially food intake and the caloric content of a meal can affect drug transit time, luminal dissolution and drug permeability. Thus, the prandial state may have a significant impact on the in vivo behaviour of such formulations as a whole and particularly on the drug bioavailability.

For GITS formulations, such as Adalat® XL®, Adalat® LA, Adalat® Crono, Adalat® OROS, earlier studies have demonstrated that no significant influence of concomitant food-intake occurs.

ELIGIBILITY:
Inclusion Criteria:

1. sex: male
2. ethnic origin: Caucasian
3. age: 18 - 55 years, inclusive
4. body-mass index (BMI): ³ 22 kg/m² and £ 27 kg/m²
5. good state of health (no clinically significant deviations from normal clinical results and laboratory findings)
6. the subject must give written informed consent, after having been informed about benefits and potential risks of the trial, as well as details of the insurance taken out to cover the subject's participating in the study

Exclusion Criteria:

1. existing cardiac or haematological diseases and/or pathological findings, which might interfere with the drug's safety, tolerability, absorption and/or pharmacokinetics
2. existing hepatic and/or renal diseases and/or pathological findings, which might interfere with the drug's safety, tolerability, absorption and/or pharmacokinetics
3. existing gastrointestinal diseases and/or pathological findings, including severe gastrointestinal or esophageal constriction or narrowing, which might interfere with the drug's safety, tolerability, absorption and/or pharmacokinetics
4. history of relevant CNS and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
5. relevant pathological changes in the ECG (12 standard leads) such as a second- or third-degree AV block, complete bundle branch block, prolongation of the QRS complex over 120 msec or the QTc-interval above 450 msec
6. known allergic or intolerance reactions to the active ingredient used or to constituents of the pharmaceutical preparations (e.g. lactose intolerance)
7. subjects with severe allergies or multiple drug allergies
8. systolic blood pressure below 110 mmHg or above 155 mmHg
9. diastolic blood pressure below 60 mmHg or above 95 mmHg
10. resting heart rate in the awake subject below 45 bpm or above 90 bpm
11. laboratory values out of normal range unless the deviation from normal is judged as not relevant for the study by the investigator
12. positive anti-HIV-test, HBs-AG-test or anti-HCV-test Lack of suitability for the trial
13. acute or chronic diseases which could affect absorption or metabolism
14. history of or current drug or alcohol dependence
15. regular intake of alcoholic food or beverages of ≥ 40 g pure ethanol per day
16. subjects who are on a diet which could affect the pharmacokinetics of the drug
17. regular intake of caffeine containing food or beverages of ≥ 500 mg (calculated as caffeine) per day
18. heavy smokers (≥ 10 cigarettes per day or equivalents of other nicotine containing products)
19. blood donation or other blood loss of more than 400 ml within the last two months prior to the start of the study
20. participation in a clinical trial during the last two months prior to individual enrolment of the subject
21. regular treatment with any systemically available medication (except hormonal replacement therapy e.g. L-thyroxine)
22. subjects, who report a frequent occurrence of migraine attacks Administrative reasons
23. subjects suspected or known not to follow instructions
24. subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to as a result of their participation in the study -

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
PK parameters after s.d. of 60 mg Nifedipine(Bayer Healthcare AG manufactured asAdalat XL,Adalat LA,Adalat Crono,Adalat OROS)and Gen-nifedipine extended release,(previously named as Gen-Nifedipine XL),administered under fasting/fed condition

SECONDARY OUTCOMES:
Descriptive characterisation of safety and tolerability of the investigational products in the study population

CONTACTS AND LOCATIONS:
Overall Officials: Frank Donath, MD, Principal Investigator — SocraTec R&D GmbH
Locations (1):
- SocraTec R&D Probandenstation, Erfurt, Thuringia, Germany